CLINICAL TRIAL: NCT01984580
Title: Effect of Zinc on Barrett's Metaplasia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Main Line Health (Other)
Collaborators: Sharpe-Strumia Research Foundation (Other)
Responsible Party: Principal Investigator, James M. Mullin, Ph.D., Professor, Main Line Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F/N-R-11-3038L
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Barrett's Metaplasia
Keywords: Barrett's esophagus; Esophagus; Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma | interventions — gluconic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zinc (Experimental)
  Interventions: Drug: zinc gluconate
- sodium (Placebo Comparator)

INTERVENTIONS:
Drug: zinc gluconate — 26.6 mg zinc BID (as zinc gluconate)
  Arms: Zinc

SUMMARY:
Using orally administered zinc to patients already diagnosed with the pre-cancerous condition, Barrett's Esophagus, this study is asking two questions:

1. can this zinc administration cause molecular-level changes in the Barrett's tissue?
2. are the changes measured indicative of chemopreventive action by zinc regarding cancer progression?

DETAILED DESCRIPTION:
14 days prior to already-scheduled upper endoscopy (EGD) procedures for routine surveillance of Barrett's tissue, patients who have given written, informed consent are randomized (sealed envelope method) and placed on an oral dose of zinc gluconate (26.6 mg zinc BID) or a placebo (molar equivalent of sodium gluconate BID) for 14 days. At the time of endoscopy, 4 biopsies are taken (and pooled) from the Barrett's tissue and 4 from proximal normal esophageal tissue. Biopsies are flash frozen for later analyses by atomic absorption spectroscopy, PAGE and Western immunoblot or RNA microarray.

ELIGIBILITY:
Inclusion Criteria:ages 18-80; prior diagnosis of Barrett's esophagus -

Exclusion Criteria:unable to provide written, informed consent; prior history of Barrett's dysplasia or esophageal adenocarcinoma; drug exclusions: hormone replacement therapy, cholestyramine, amiloride diuretics, oral quinolone antibiotics, glucocorticoids, corticosteroids, anticoagulants (other than aspirin)

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-04; Primary Completion 2015-03 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Changes in zinc-regulated cellular proteins within Barrett's tissue | in biopsy tissue after 14 days of Zn exposure

SECONDARY OUTCOMES:
Changes in cellular microRNA profile; changes in protein cancer biomarkers | in biopsy tissue after 14 days of Zn exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Lankenau Institute for Medical Research, Wynnewood, Pennsylvania, United States